CLINICAL TRIAL: NCT06330597
Title: Noninvasive Versus Invasive Assessment of Hemodynamics in the Cardiac Intensive Care Unit
Brief Title: NIVIA-Hemodynamics
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-5196
Record Dates: First submitted 2022-05-30; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Cardiogenic Shock; Heart Failure; Shock; Hemodynamic Instability
Keywords: Pulmonary Artery Catheter; Lung Ultrasound; Echocardiography
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure; Shock | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to CICU: The study population will be composed of patients admitted to the Coronary Intensive Care Unit (CICU) requiring hemodynamic assessment using pulmonary artery catheter (PAC) as standard of care.
  Interventions: Diagnostic Test: Echocardiography and lung ultrasound

INTERVENTIONS:
Diagnostic Test: Echocardiography and lung ultrasound — All patients will undergo non-invasive echocardiogram and lung ultrasound at times of assessment of hemodynamic parameters as needed by usual clinical management.

SUMMARY:
This is an investigator-initiated, single-center, single-arm prospective study to compare non-invasive hemodynamic assessment using transthoracic echocardiography (TTE) and lung ultrasound (LUS) and hemodynamic assessment using PAC. Patients who have been hemodynamically assessed using PAC will be invited to participate. Each patient will undergo TTE and LUS immediately after first invasive assessment, and again daily after PAC assessments.

DETAILED DESCRIPTION:
Background

Heart Failure

Approximately 600,000 Canadians are living with heart failure (HF) with 50,000 new patients diagnosed each year. Once diagnosed, the median survival for HF patients is 1.7 years for men and 3.2 years for women. As HF progresses, patients experience a worsening in symptom severity, functional capacity, and quality of life. In addition, acute exacerbations of HF is the most frequent cause of unscheduled hospital admissions. Almost 83% of all HF patients will be hospitalized at least once and 43% hospitalized more than three times. However, the mechanisms of HF decompensation are still unclear.

Most drugs (ACE-I/ARB/beta-blockers/MRA) used for the treatment of HF are prescribed because of their ability to improve symptoms or survival. The target doses of these drugs are generally selected on the basis of reported results from randomized controlled trials rather than changes produced in cardiac monitoring of hemodynamics. Interestingly, hemodynamic monitoring has been reportedly indicated in patients where it is difficult to determine their volume status, in addition to those patients refractory to therapy. The ACC/AHA 2013 guidelines3 define the importance of invasive hemodynamic monitoring in patients with:

* severe clinical decompensation in which therapy is limited by elevated filling pressures, hypoperfusion, and vascular tone
* persistent severe symptoms despite a trial of recommended therapies
* the needed or dependency for (or escalation of) pressor and inotropic therapy

Cardiogenic shock

Cardiogenic shock (CS) is a state of profound HF resulting in peripheral organ hypoperfusion, injury and failure. The precipitating events leading to CS are diverse. Patients may experience CS as a slow progression of chronic HF. More frequently however; patients experience CS after an acute cardiac insult such as an acute myocardial infarction, myocarditis or malignant ventricular arrhythmia. It is inevitable that patients who develop CS will die if treatment is not initiated rapidly. In addition, if initial medical therapy fails to maintain adequate cardiac output, initiation of mechanical circulatory support (MCS) represents a life-saving strategy. There has been no established role for the use of invasive hemodynamic measurements in the management of patients with HF. And yet, patients with CS being considered for cardiac transplantation or placement of an MCS device are required to undergo right-heart catheterization using pulmonary artery catheter (PAC), including an assessment of right heart filling pressures, pulmonary artery pressures, left heart filling pressures and cardiac output.

University Health Network (UHN) has the largest and most comprehensive MCS program in Canada. As clinicians working at the Peter Munk Cardiac Centre (PMCC) we are caring for an ever-increasing number of patients with profound refractory cardiogenic shock who require invasive hemodynamic assessment.

Rationale for the study

The majority of patients who present to the CICU require invasive hemodynamic assessment as part of their usual care. To assist in the management of these critically ill patients, the investigators need a complete understanding of the hemodynamic status. Currently, this is usually done invasively by placing a PAC. Alternatively, a non-invasive assessment using transthoracic echocardiography (TTE) can be pursued.

Pulmonary artery Catheter

In early retrospective registries, there was no benefit shown for the use of PAC. However, this had not been studied in patients with CS until recently. In a large retrospective study of CS patients, the use of PAC was associated with improved survival (30% vs 38%). This study provided the basis for the incorporation of PAC into CS treatment algorithms. In addition, the guidelines and scientific statements limited recommendations regarding PAC to use in patients with CS. The hemodynamic data obtained with a PAC can facilitate clinical decision-making and allow customization of a treatment plan through the optimization of medical therapy. However, as with any invasive diagnostic tool, the benefit must be balanced against risks. Complications of PAC include central venous access-related adverse events (<3.6%), arrhythmias and heart block (0.3% to 3.8%), and pulmonary artery rupture (0.02% to 0.03%).

Transthoracic echocardiography

TTE is a non-invasive ultrasound-based diagnostic tool that has the ability to also evaluate and track both RV and LV hemodynamic status. There is conflicting evidence of the utility of TTE monitoring in reflecting the hemodynamic changes in PAC-derived hemodynamic measurements.

Lung Ultrasound (LUS)

LUS allows for a rapid point-of-care evaluation of a number of conditions, including pulmonary edema, lung consolidation, pleural effusion, and pneumothorax. High intra-rater and inter-rater reproducibility, ease of learning, short exam duration (<5 min), and the noninvasive nature of this technique makes it an advantageous point-of-care tool. LUS is increasingly used in the acute care setting, and has improved diagnostic accuracy compared with clinical assessment and chest radiography for the identification of a cardiac aetiology in patients presenting to the emergency department with undifferentiated dyspnea. Quantification of B-lines (vertical artefacts that result from an increase in interstitial density) has been shown to be useful for the diagnosis, monitoring, and risk assessment of patients with known or suspected ADHF. Either curvilinear or phased array transducers can be used, typically at an imaging depth of 14-18 cm.

Hypothesis

The investigators hypothesize that non-invasive hemodynamic parameters derived from TTE would be comparable to those obtained invasively by PAC in patient admitted to the CICU. The investigators also hypothesize that there will be a strong correlation between intracardiac pressures and the severity of pulmonary congestion as evaluated by LUS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with admitted to the CICU in whom PAC is inserted as standard of care,

Exclusion Criteria:

* Enrollment into another trial with an active treatment arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of patients admitted to the Coronary Intensive Care Unit (CICU) requiring hemodynamic assessment using pulmonary artery catheter (PAC) as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-17 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between E/e' ratio and PCWP vs. correlation between lung ultrasound score and PCWP. | Day 1
  To determine whether non-invasive assessment of hemodynamics by echocardiogram are comparable to invasive measurements.

SECONDARY OUTCOMES:
Correlation between cardiac output measured by echocardiography (using LVOT diameter and VTI) and by PAC (using thermodilution) | Day 1, Day 2
  To correlate cardiac and pulmonary pressures derived from invasive measurements with lung ultrasound findings.
Correlation between right atrial pressure assessed by echocardiography (using IVC diameter and respiratory variation) and by PAC | Day 1, Day 2
  To correlate cardiac and pulmonary pressures derived from invasive measurements with lung ultrasound findings.
Correlation between pulmonary pressure assessed by echocardiography (using TR max velocity and estimated RAP) and by PAC | Day 1, Day 2
  To correlate cardiac and pulmonary pressures derived from invasive measurements with lung ultrasound findings.
Correlation between pulmonary pressure assessed by echocardiography (using PAT) and by PAC | Day 1, Day 2
  To correlate cardiac and pulmonary pressures derived from invasive measurements with lung ultrasound findings.
Correlation between PVR assessed by echocardiography (using PAT) and by PAC | Day 1, Day 2
  To correlate cardiac and pulmonary pressures derived from invasive measurements with lung ultrasound findings.
Correlation between right ventricular function assessed by echocardiography (using TAPSE and S') and by PAC (using PAPI and RVSWI) | Day 1, Day 2
  To correlate cardiac and pulmonary pressures derived from invasive measurements with lung ultrasound findings.
Correlation between E/e' ratio and PCWP vs. correlation between lung ultrasound score and PCWP. | Day 2
  To determine whether non-invasive assessment of hemodynamics by echocardiogram are comparable to invasive measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Filio Billia, MD PhD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No